CLINICAL TRIAL: NCT03192553
Title: Alternative Doffing Strategies to Prevent Healthcare Worker Self-Contamination When Using Personal Protective Equipment (PPE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20009234
Record Dates: First submitted 2017-05-26; First posted 2017-06-20 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Personal Protective Equipment
Keywords: donning; doffing; self-contamination; healthcare workers

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a doffing protocol chronologically starting with the double glove and ending with the control until 100 volunteers have participated. Only one volunteer with participate in each simulation session.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Double Gloving Procedure (Experimental): Participants will doff PPE using a double gloving procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Interventions: Behavioral: Double Gloving Procedure
- Intensified Hand Hygiene Procedure (Experimental): Participants will doff PPE using an intensified hand hygiene procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Interventions: Behavioral: Intensified Hand Hygiene Procedure
- One-Step Procedure (Experimental): Participants will doff PPE using a one-step procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Interventions: Behavioral: One Step Procedure
- CDC Procedure (Control) (Other): Participants will doff PPE following the CDC procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Interventions: Behavioral: CDC Procedure

INTERVENTIONS:
Behavioral: Double Gloving Procedure — Participants will doff PPE using a double gloving procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Arms: Double Gloving Procedure
Behavioral: Intensified Hand Hygiene Procedure — Participants will doff PPE using an intensified hand hygiene procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Arms: Intensified Hand Hygiene Procedure
Behavioral: One Step Procedure — Participants will doff PPE using a one-step procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Arms: One-Step Procedure
Behavioral: CDC Procedure — Participants will doff PPE using a CDC recommended procedure after coating with Glogerm fluorescent dye +/- staphylococcus epidermidis
  Arms: CDC Procedure (Control)

SUMMARY:
Alternative doffing strategies may help prevent self-contamination of staff members when using PPE. The study aims to determine which among the suggested methods in the literature that have been proposed as alternatives to the traditional CDC recommended doffing protocol, would be most beneficial to reduce healthcare worker self-contamination.

DETAILED DESCRIPTION:
A randomized controlled trial of doffing procedures will be conducted by healthcare worker volunteers who participate in direct patient care. However, doffing simulations will be conducted outside of patient care areas and will not involve patients. Staff participants PPE techniques will be evaluated in the controlled environment of the simulation center of the Unique Pathogens Unit. The comparison groups will be the Centers for Disease Control (CDC) procedure with the addition of a second layer of gloves (double gloving procedure), the CDC procedure with additional hand hygiene performed on gloves at key steps (intensified hand hygiene procedure), and the one-step roll off of gown and gloves (one-step procedure), with the CDC procedure as the control. Participants will be assigned to a doffing protocol chronologically starting with the double glove and ending with the control until 100 volunteers have participated. Additional PPE such as masks and goggles will be removed as part of each of the four protocols. Healthcare workers will receive a demonstration of the donning/doffing from the study coordinator, and perform a practice donn/doff prior to the observed simulation. Only one volunteer with participate in each simulation session. Glogerm (TM) will be applied to PPE in a thin stripe and smoothed to evenly with gloved hands to cover arms, trunk, and gown hem. S. epidermidis will be applied using colonies diluted in solution and spread over gloves, arms, trunk, hem with a swab.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Providers at VCU Medical Center, including medical degree holding trainees who are medical housestaff Adults > or =18 years of age

Exclusion Criteria:

students pregnant or breastfeeding healthcare workers non-clinical providers children/teens <18 years of age open skin lesions or dermatitis presence of prosthetic materials such as prosthetic joints, heart valves

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Self-contamination rate | Assessed immediately after each post-doffing simulation - self-contamination will be documented during the simulation appointment, immediately following doffing, by visual assessment
  Measure of frequency of contamination by body site for each doffing procedure via visual assessment

SECONDARY OUTCOMES:
Acceptability of doffing procedure to healthcare workers | Assessed immediately after each post-doffing simulation - the questionnaire will be administered before the participant leaves the simulation appointment
  Aspects of acceptability such as ease, comfort, and efficacy measured by Likert Scale Staff Questionnaire (1=strongly disagree, 5=strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Doll, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States